CLINICAL TRIAL: NCT04771364
Title: Impact of "ASAP" Multidisciplinary Optimization Care Protocol on Clinical Outcome in Elderly Inpatients for Hip Fracture: Retrospective Cohort Study
Brief Title: Impact of "ASAP" Multidisciplinary Optimization Care Protocol on Clinical Outcome in Elderly Inpatients for Hip Fracture
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Head of Anesthesiology Departement, University of Liege
Other Study IDs: ASAP
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard care: Patients aged >65 years old scheduled for hip fracture between January 1st 2017 and December 31th 2019.
  Standard anesthesiology cares were performed, as usual in our hospital institution.
- ASAP cohort: Patients aged >65 years old scheduled for hip fracture between January 1st 2020 and December 31th 2022.
  Standard anesthesiology cares were performed, as usual in our hospital institution, but the investigator focused the attention on these cares' adaptation: early geriatrician's advice, prefer locoregional anesthesia techniques where possible, early surgical therapy and medical adaptation on chronic therapy.
  Interventions: Other: ASAP care's protocol

INTERVENTIONS:
Other: ASAP care's protocol — Early geriatrician's advice, prefer locoregional anesthesia techniques where possible, early surgical therapy and medical adaptation on chronic patient's therapy (in particular with regard to sedative, anticholinergic and psychotropic drugs).
  Groups: ASAP cohort

SUMMARY:
To compare the impact of ASAP protocol (geriatric advice, early surgery, loco-regional anesthesia and pharmacological adaptation) on elderly patients with hip fracture and clinical outcome.

DETAILED DESCRIPTION:
Retrospective double cohort analysis for ASA physical status 1, 2 and 3 elderly patients >65 years old, scheduled to undergo surgery for hip fracture between January 1st 2017 and December 31st 2022.

The investigator want to confirm the better outcome on 30-days mortality after surgery in patients where the ASAP protocol was applied, starting from 1 January 2020.

ASAP protocol follow the latest international guidelines about hip fracture in elderly patient. The investigator focuses the research about the impact of ASAP protocol on clinical outcome: geriatrician's advice, impact of loco-regional techniques on intra-operative and postoperative pain control, chronic pharmacological therapy's adaptation and 30-days postoperative mortality.

ELIGIBILITY:
Inclusion Criteria:

* Over 65 years old patients with hip fractures between January 1st 2017 and December 31th 2022

Exclusion Criteria:

* Fracture without indication for surgery
* Death before surgery
* Intensive care's or polytrauma patients (> 2 fracture sites) or under pharmacological coma needed before and after surgery.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients >65 years old with hip fracture
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 7 days
  Neurological, cardiovascular, pulmonary, renal, infectious and gastrointestinal complications after surgery.

SECONDARY OUTCOMES:
Days of hospitalisation | 30 days
  Total hospitalisation days
30-days postoperative mortality | 30 days
  Mortality 1 month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borges FK, Bhandari M, Patel A, Avram V, Guerra-Farfan E, Sigamani A, Umer M, Tiboni M, Adili A, Neary J, Tandon V, Sancheti PK, Lawendy A, Jenkinson R, Ramokgopa M, Biccard BM, Szczeklik W, Wang CY, Landoni G, Forget P, Popova E, Wood G, Nabi Nur A, John B, Sleczka P, Feibel RJ, Balaguer-Castro M, Deheshi B, Winemaker M, de Beer J, Kolesar R, Teixidor-Serra J, Tomas-Hernandez J, McGillion M, Shanthanna H, Moppett I, Vincent J, Pettit S, Harvey V, Gauthier L, Alvarado K, Devereaux PJ. Rationale and design of the HIP fracture Accelerated surgical TreaTment And Care tracK (HIP ATTACK) Trial: a protocol for an international randomised controlled trial evaluating early surgery for hip fracture patients. BMJ Open. 2019 May 1;9(4):e028537. doi: 10.1136/bmjopen-2018-028537. PMID 31048449
- [Result] Matsuo M, Yamagami T, Higuchi A. Impact of age on postoperative complication rates among elderly patients with hip fracture: a retrospective matched study. J Anesth. 2018 Jun;32(3):452-456. doi: 10.1007/s00540-018-2494-8. Epub 2018 Apr 16. PMID 29663067